CLINICAL TRIAL: NCT02283515
Title: Efficacy of Locally Delivered 1.2% Rosuvastatin Gel in Non Surgical Treatment of Chronic Periodontitis Patients: A Randomised Clinical Control Trial.
Brief Title: Efficacy of Locally Delivred 1.2% Rosuvastatin Gel in Chronic Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Proffesor and Head, dept of periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/10/2013-14A
Record Dates: First submitted 2014-09-27; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Periodontitis
Keywords: chronic periodontitis; local drug delivery; rosuvastatin; osseo-differentiation
MeSH Terms: conditions — Chronic Periodontitis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group I - Rosuvastatin, 1.2 mg (Active Comparator): Rosuvastatin- locally placed in intrabony defect sites.
  Interventions: Drug: Rosuvastatin
- group II - placebo (Placebo Comparator): placebo-placed locally in intrabony defects.

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin (RSV) is one of new synthetic, second-generation, sulfur-containing, hydrophilic statin, a highly efficient competitive inhibitors of HMG CoA Reductase having important role in reducing serum cholesterol concentrations and lowers the risk of cardiovascular disease.
  Other Names: Hydrophilic statin
  Arms: group I - Rosuvastatin, 1.2 mg

SUMMARY:
BACKGROUND: Chronic periodontitis (CP) is an inflammatory condition affecting tooth supporting tissues and alveolar bone that surround the tooth leading to formation of deepend gingival sulcus that is highly prone to pathologic changes, ultimately bone resorption and tooth loss. In the literature, several pharmacologic agents have been administration via local delivery route, directly into diseased sites affirming greater improvement in periodontal status. Therefore, present study was conducted to determine the clinical effectiveness of subgingivally delivered 1.2% Rosuvastatin gel incorporated into an methylcellulose vehicle for its controlled release into intrabony defect sites in adjunct to scaling and root planing for treatment of chronic periodontitis patients.

MATERIAL AND METHODS: Sixty five patients were categorized into two treatment groups: group I -SRP plus RSV, 1.2 mg and group II -SRP plus placebo. Clinical parameters included modified sulcus bleeding index (mSBI), probing depth (PD), and clinical attachment level (CAL), were recorded at baseline before SRP and at 1, 3, 4, and 6 months. Radiologic assessment of intrabony defect (IBD) fill was analysed at baseline and after 6months using computer-aided software.

DETAILED DESCRIPTION:
Rosuvastatin (RSV) is one of new synthetic, second-generation, sulfur-containing, hydrophilic statin, a highly efficient competitive inhibitors of HMG CoA Reductase having important role in reducing serum cholesterol concentrations and lowers the risk of cardiovascular disease. It has potent anti-inflammatory effects, mediated via vascular endothelium derived nitric oxide (eNO) that inhibits P selectin synthesis by endothelial cells. This protective action is evidenced by reduced levels of high-sensitivity C-Reactive Protein (hs-CRP) , a clinical marker of inflammation produced in response to proinflammatory cytokines such as interleukin-6 (IL-6), therefore it contributes to the prevention and remission of inflammatory diseases. Recently, an in-vivo study demonstrated that RSV promotes osteoblast differentiation, by regulating the expression of solute carrier (Slco1a1), which may constitute the transport system for RSV across the cell membrane in mature osteoblasts.

SRP plus RSV(1.2 mg/0.1 ml) in situ gel (group I) or SRP plus placebo gel (group II) local drug delivery

ELIGIBILITY:
Inclusion Criteria:

* Systemically sound with moderate probing depth (PD) of 5- 6 mm or clinical attachment loss (CAL) of 4 - 6 mm) or deep pockets (PD ≥ 7 mm or CAL of 6 - 9 mm) and vertical bone loss ≥ 3 mm on intraoral periapical radiographs.
* Subjects with ≥ 20 teeth with no history of periodontal therapy in the preceding 6 months nor under any antibiotic therapy were included in the study.

Exclusion Criteria:

* Patients on systemic statin therapy with known or suspected allergy to the RSV group, patients with any other forms of periodontitis, use of tobacoo in any form, smokers, alcoholics, immune-compromised and systemically unhealthy patients, and pregnant or lactating females were excluded.

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study was complete bone defect fill. | 24 weeks complete bone defect fill.
  Using radiographic analyser bone defect fill was analysed

SECONDARY OUTCOMES:
Probing Depth. | an average of 24 weeks Probing depth
  Using UNC-15 probe
Clinical Attachment Level | 24 weeks
  Using UNC-15 probe and acrylic stents CAL was analysed
modified Sulcus BIeeding Index | 12 and 24 weeks
  Using a WALKING METHOD OF PROBING